CLINICAL TRIAL: NCT06041126
Title: The Effect of Disease Severity and Respiratory Functions on Muscle Oxygenation in Stable COPD Patients
Brief Title: The Effect of Clinical Parameters on Muscle Oxygenation in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Gulhan Yilmaz Gokmen, Assistant Professor, Bandırma Onyedi Eylül University
Other Study IDs: 2023-72
Record Dates: First submitted 2023-04-27; First posted 2023-09-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Muscle Oxygenation; Disease Severity; Respiratory Function
Keywords: Chronic Obstructive Pulmonary Disease; Muscle Oxygenation; Disease Severity; Respiratory Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group one: Patients with COPD according to the combined COPD assessment Global Intervention (GOLD) guidelines, participants who are in groups A and B (mild-moderate) will be included in group 1.
- Group two: COPD patients according to the combined COPD assessment, according to the "Global Intervention (GOLD) guidelines", participants who are in groups C and D (severe-very severe) will be included in group 2.

SUMMARY:
The aim of this study is to examine the peripheral muscle oxygenation of patients with Chronic Obstructive Pulmonary Disease at rest, during submaximal exercise and recovery, and to examine the effects of disease severity and respiratory functions on peripheral muscle oxygenations. In this study, the effect of disease severity and respiratory problems on peripheral muscle metabolism of patients with COPD will be explained.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD (according to GOLD Staging: GOLD 1, GOLD 2, GOLD 3, GOLD 4)
* Being between the ages of 40-80
* Body Mass Index <35
* Not having an acute exacerbation in the last 3 months

Exclusion Criteria:

* Patients who do not want to participate in the study
* Arthritis causing weakness in the lower extremity, neurological disease, deep vein thrombosis, peripheral arterial disease, muscle weakness, fracture etc. patients with the condition
* Common diseases such as malignancy, pulmonary embolism, vasculitis, collagen tissue diseases, interstitial fibrosis, severe pneumonia patients with parenchymal destruction
* Patients with severe dyspnea and hemodynamic instability who cannot perform the 6 Minute Walk Test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable COPD Patients
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Muscle oxygenation | one day
  The muscle oxygen monitor is a lightweight (42 g) and small (dimensions: 61 × 44 × 21

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale | one day
  Medical Research Council (MRC) Dyspnea Scale will be used to assess the severity of dyspnea. The severity of dyspnea during activities of daily living is graded from 0 to 4 on the Medical Research Council (MRC) Dyspnea Scale.
COPD Assessment Test (CAT) | one day
  The COPD Assessment Test (CAT) is a new scoring system for COPD patients, which provides a simple method for assessing the impact of COPD on the patient's health. Range of CAT scores from 0-40.
Charlson Comorbidity Index | one day
  The Charlson Comorbidity Index was first developed in 1987 by Mary Charlson and colleagues as a weighted index to predict risk of death within 1 year of hospitalization for patients with specific comorbid conditions. Nineteen conditions were included in the index. The total score in the CCI is derived by summing the assigned weights of all comorbid conditions presented by the client. Higher scores indicate a more severe condition and consequently, a worse prognosis.
Quadriceps muscle strength measurement | one day
  Quadriceps muscle strength measurement of the patients will be evaluated with a manual muscle strength measuring device (Lafayette Instrument, USA) and recorded in kg/force. In muscle strength measurements, maximal voluntary isometric contraction (make test), which is reported to be more reliable in the literature and is frequently used, will be used. It will be repeated three times in both lower extremities with an interval of 30 seconds and the highest measurement will be recorded. For quadriceps muscle strength measurement, the patients will be seated on the treatment table with their legs hanging down and the thigh will be fixed by placing a rolled towel under the knee joint of the side to be evaluated. In this position, the patient will be asked to extend until the knee is locked, and the resistance will be given just above the ankle joint.
Six-minute walking test | one day
  It is a submaximal exercise capacity measurement test. The patient is asked to walk as briskly as possible on a flat surface of 30 meters for 6 minutes. In our study, the test will be carried out in a 30-meter corridor in accordance with the guidelines.
Pulmonary Function Test | one day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria.
Maximum Inspiratory Pressure / Maximum Expiratory Pressure Measurement | one day
  Respiratory muscle strength of individuals will be measured using an electronic and portable oral pressure measurement device, according to ATS / ERS criteria, with COSMED brand Pony FX model portable spirometer (COSMED, Italy). It is one of the most commonly used and noninvasive methods for the evaluation of respiratory muscle strength. With this method, maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) are measured. MIP and MEP are intraoral pressures measured during maximal breathing against a valve that closes the airway during maximal inspiration and expiration.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No